CLINICAL TRIAL: NCT03238781
Title: A Phase 2a Randomized Double-blind Placebo Controlled Study to Evaluate the Efficacy and Safety of AMG 301 in Migraine Prevention
Brief Title: Study to Evaluate the Efficacy and Safety of AMG 301 in Migraine Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20150308; 2017-000630-57 (EudraCT Number)
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Chronic Migraine or Episodic Migraine
Keywords: Migraine; Headache; Prevention; Prophylaxis
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants randomized to Placebo were administered 6 subcutaneous (SC) injections on day 1 and weeks 2, 4, 6, 8 and 10 during the 12 week double-blind treatment period.
  Interventions: Drug: Placebo
- AMG 301 210 mg Q4W (Experimental): Participants randomized to AMG 301 210 mg every fourth week (Q4W) received a total of 3 AMG 301 subcutaneous (SC) injections (70 mg/mL in each injection) plus 3 matching placebo injections on day 1 and weeks 4 and 8. Participants also received 6 SC placebo injections on weeks 2, 6, and 10 during the 12 week double-blind treatment period.
  Interventions: Drug: AMG 301
- AMG 301 420 mg Q2W (Experimental): Participants randomized to AMG 301 420 mg every second week (Q2W) received a total of 6 AMG 301 subcutaneous (SC) injections (70 mg/mL in each injection) on day 1 and weeks 2, 4, 6, 8, and 10 during the 12 week double-blind treatment period.
  Interventions: Drug: AMG 301

INTERVENTIONS:
Drug: Placebo — Placebo was presented in identical containers, stored/packaged the same as AMG 301. All injections were administered within 30 minutes on treatment days.
  Arms: Placebo
Drug: AMG 301 — AMG 301 was packaged in 5 mL clear glass vials containing 1 mL of 70 mg/mL of AMG 301. All injections were administered within 30 minutes on treatment days.
  Arms: AMG 301 210 mg Q4W; AMG 301 420 mg Q2W

SUMMARY:
To evaluate the effect of AMG 301 compared to placebo on the change from the baseline period in monthly migraine days in subjects with migraine.

DETAILED DESCRIPTION:
A Phase 2a, randomized, double-blind, placebo-controlled, 3-arm parallel group study to evaluate the efficacy and safety of AMG 301 in subjects with chronic migraine or episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 to ≤ 60 years of age at the time of signing the informed consent form.
* History of migraine (with or without aura) for ≥ 12 months before screening according to the International Headache Society (IHS) Classification ICHD-III (Headache Classification Committee of the International Headache Society, 2013)
* Migraine frequency: ≥ 4 migraine days per month on average across the 3 months before screening.
* Failed at least 1 medication for prophylactic treatment of migraine due to tolerability or lack of efficacy

Exclusion Criteria:

* Older than 50 years of age at migraine onset.
* History of cluster headache, hemiplegic migraine headache.
* Unable to differentiate migraine from other headaches.
* Migraine with continuous pain, in which the subject does not experience any pain-free periods (of any duration) during the 1 month before the screening period.
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 343 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (45):
- United States (21):
  - Research Site, Long Beach, California
  - Research Site, Santa Monica, California
  - Research Site, Boulder, Colorado
  - Research Site, East Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, City of Saint Peters, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Plainview, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Vienna
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Markham, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Prague
  - Research Site, Přerov
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Glostrup Municipality
  - Research Site, Viborg
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Oulu
  - Research Site, Turku
- Germany (4):
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Leipzig
- Research Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Ashina M, Dolezil D, Bonner JH, Zhou L, Klatt J, Picard H, Mikol DD. A phase 2, randomized, double-blind, placebo-controlled trial of AMG 301, a pituitary adenylate cyclase-activating polypeptide PAC1 receptor monoclonal antibody for migraine prevention. Cephalalgia. 2021 Jan;41(1):33-44. doi: 10.1177/0333102420970889. Epub 2020 Nov 24. PMID 33231489
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 510 subjects were screened.
Pre-assignment Details: Participants were randomized 4:3:3 to placebo, AMG 301 210 mg Q4W, or AMG 301 420 mg Q2W, respectively. The randomization was stratified by
  * chronic migraine versus episodic migraine and
  * North America versus Rest of World.
Period: Overall Study
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Started | 137 | 104 | 102
Completed | 111 | 87 | 82
Not Completed | 26 | 17 | 20
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Withdrawal by Subject | 23 | 14 | 16
Not completed — Decision by sponsor | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set consisting of participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W | Total
Number analyzed (Participants) | 137 | 104 | 102 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (9.9) | 42.3 (9.7) | 42.5 (9.4) | 42.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 94 | 90 | 301
  Male | 20 | 10 | 12 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 3 | 15
  Not Hispanic or Latino | 131 | 98 | 99 | 328
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 4 | 12
  White | 129 | 100 | 96 | 325
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 71.8 (15.0) | 73.8 (17.2) | 72.1 (14.9) | 72.5 (15.7)
Height [Mean (Standard Deviation); unit: cm] | 168.27 (7.82) | 167.05 (8.56) | 167.55 (7.72) | 167.69 (8.01)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.29 (4.66) | 26.37 (5.45) | 25.64 (4.78) | 25.72 (4.95)
Monthly Migraine Days [Mean (Standard Deviation); unit: monthly migraine days] — A migraine day is any calendar day from the eDiary in which the participant experienced a migraine headache. A migraine headache is a headache with or without aura, lasting for >= 4 hours, and meeting >=1 of the criteria:
  1. >= 2 pain features (unilateral, throbbing, moderate to severe, exacerbated with exercise/physical activity)
  2. >= 1 symptoms (nausea and/or vomiting, photophobia and phonophobia) If the participant took a migraine-specific medication during aura or to treat headache, it was counted as a migraine day. Baseline timeframe was the 28-day period prior to study treatment.
  monthly migraine days | 12.18 (5.14) | 12.47 (4.78) | 12.14 (5.32) | 12.26 (5.08)
Monthly Headache Days [Mean (Standard Deviation); unit: days] — A headache day is any calendar day from the eDiary in which the participant experiences a headache (initial onset, continuation or recurrence of the headache). A qualified headache is defined as:
  * a migraine headache (including an aura-only event that is treated with acute migraine-specific medication), or
  * a non-migraine headache, which is a headache that lasts >= 4 hours and is not a migraine headache, or
  * a headache of any duration for which acute headache treatment is administered. Baseline timeframe was the 28-day period prior to study treatment.
  days | 13.45 (5.27) | 13.85 (4.90) | 13.09 (5.24) | 13.46 (5.15)
Targeted Neurological Disease Diagnosis [Number; unit: participants with diagnosis] — Each participant may contribute to more than one category
  participants with diagnosis
    Migraine with aura | 40 | 32 | 43 | 115
    Migraine without aura | 120 | 92 | 87 | 299
    Depression | 24 | 25 | 18 | 67
    Anxiety | 21 | 15 | 16 | 52
Reported Reasons for Prior Migraine Prophylactic Medication Failure [Number; unit: participants reporting the reason] — Each participant may contribute to more than one category
  participants reporting the reason
    Lack of efficacy | 110 | 88 | 77 | 275
    Intolerance | 62 | 47 | 52 | 161
Baseline Migraine Type [Count of Participants; unit: Participants] — Chronic migraine (CM) was defined as:
  >= 15 headache days of which >= 8 headache days meet criteria as igraine days during the baseline period based on the electronic diary (eDiary) calculations.
  Episodic migraine was defined as:
  <15 headache days of which >=4 headache days meet criteria as migraine days during the baseline period based on the eDiary calculations.
  Participants
    Chronic migraine | 44 | 39 | 36 | 119
    Episodic migraine | 93 | 65 | 66 | 224

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days to the Last 4 Weeks of the 12 Week Double-Blind Treatment Period
Description: A migraine day is any calendar day from the eDiary in which the participant experienced a migraine headache. A migraine headache is a headache with or without aura, lasting for >= 4 hours, and meeting >=1 of the criteria:
  1. >= 2 pain features (unilateral, throbbing, moderate to severe, exacerbated with exercise/physical activity)
  2. >= 1 symptoms (nausea and/or vomiting, photophobia and phonophobia) If the participant took a migraine-specific medication during aura or to treat headache, it was counted as a migraine day.
  Days without eDiary data in each monthly interval are handled by proration.
  Negative change from baseline values indicated improvement (i.e. fewer migraine days after treatment as compared to baseline).
Time Frame: Baseline Day -28 to Day -1; Weeks 9-12
Population: Efficacy Analysis set consisting of participants who were randomized, received >=1 dose of investigational product, and have >=1 postbaseline monthly eDiary measurement. Participants were analyzed according to their randomized treatment group, regardless of treatment received.
  Participants with both baseline and week 9-12 values are included.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 119 | 93 | 85
days | -2.45 (0.40) | -2.20 (0.45) | -2.19 (0.46)
Statistical Analysis 1: Comparison: Placebo vs AMG 301 210 mg Q4W; An adjusted analysis is presented that utilized a generalized linear mixed model which included treatment, visit, treatment-by-visit interaction, stratification factors of region and baseline migraine frequency (chronic migraine vs episodic migraine), and baseline value as covariates and assuming a first-order autoregressive covariance structure. The p-values for pairwise comparisons versus placebo are nominal p-values without multiplicity adjustment; Test type: Superiority; p = 0.66, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = 0.26, 95% CI 2-sided [-0.88 to 1.40]
Statistical Analysis 2: Comparison: Placebo vs AMG 301 420 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.65, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = 0.27, 95% CI 2-sided [-0.89 to 1.43]

2. Secondary Outcome: Percentage of Participants Who Responded, Defined as At Least a 50% Reduction From the Baseline Period in Monthly Migraine Days in the Last 4 Weeks of the 12-Week Double-Blind Treatment Period
Description: Responders are participants who had at least a 50% reduction from baseline in monthly migraine days during the last 4 weeks of treatment in the 12-week double blind period.
Time Frame: Baseline Day -28 to Day -1; Weeks 9-12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 119 | 93 | 85
percentage of participants | 22.7 | 19.4 | 18.8
Statistical Analysis 1: Comparison: Placebo vs AMG 301 210 mg Q4W; The common odds ratios and p-values are obtained from a Cochran-Mantel-Haenszel test, stratified by stratification factors of region and baseline migraine frequency (chronic migraine vs episodic migraine); Test type: Superiority; p = 0.57, Cochran-Mantel-Haenszel — 2-sided significance level of 0.05; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.41 to 1.62]
Statistical Analysis 2: Comparison: Placebo vs AMG 301 420 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.45, Cochran-Mantel-Haenszel — 2-sided significance level of 0.05; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.37 to 1.54]

3. Secondary Outcome: Change From Baseline Period in Monthly Acute Migraine-Specific Medication Days in the Last 4 Weeks of the 12-Week Double-Blind Treatment Period
Description: Number of days on which acute headache medications (triptans and ergotamine-derivatives, alone or in combination) are used as recorded in eDiary. Monthly acute headache medication treatment days at baseline are the number of acute headache medication treatment days in the baseline period. Days without eDiary data are handled by proration.
  Negative change from baseline values indicate improvement (i.e. fewer days requiring acute migraine-specific medications after treatment as compared to baseline).
Time Frame: Baseline Day -28 to Day -1; Weeks 9-12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 103 | 84 | 76
days | -1.25 (0.29) | -1.28 (0.33) | -1.34 (0.34)
Statistical Analysis 1: Comparison: Placebo vs AMG 301 210 mg Q4W; Adjusted analysis utilizes a generalized linear mixed model which includes treatment, visit, treatment-by-visit interaction, stratification factors of region and baseline migraine frequency (CM versus EM), and baseline value as covariates and assuming a first-order autoregressive covariance structure. The p-values for pairwise comparisons versus placebo are nominal p-values without multiplicity adjustment; Test type: Superiority; p = 0.94, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = -0.03, 95% CI 2-sided [-0.87 to 0.81]
Statistical Analysis 2: Comparison: Placebo vs AMG 301 420 mg Q2W; Test type: Superiority; p = 0.84, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = -0.09, 95% CI 2-sided [-0.94 to 0.77]

4. Secondary Outcome: Change From Baseline in Mean Physical Impairment Domain Scores as Measured by the Migraine Physical Function Impact Diary (MPFID) Over the Last 4 Weeks of the 12-Week Double-Blind Treatment Period
Description: Participants complete the MPFID every day during baseline (Days -28 to Day -1) and the 12-week Double Blind Treatment Period. The MPFID has 2 domains, Impact on Everyday Activities (7 items) and Physical Impairment (5 items), and 1 stand-alone global question that provides an assessment of the overall impact of migraine on participants' everyday activities. The recall period for each item is the past 24 hours.
  The Physical Impairment Domain Score is reported here. A participant's response to the difficulty of the 5 physical impairment items is measured using a 5-point scale, with difficulty measurements ranging from 1 to 5. The sum was rescaled to a 0 to 100 scale, with 0=no difficulty and 100=unable to do (maximum burden). Negative change from baseline values indicate improvement in migraine impact.
Time Frame: Baseline Day -28 to Day -1; Weeks 9-12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 119 | 93 | 85
units on a scale | -2.44 (0.78) | -2.72 (0.89) | -2.13 (0.91)
Statistical Analysis 1: Comparison: Placebo vs AMG 301 210 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.81, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = -0.28, 95% CI 2-sided [-2.56 to 2.01]
Statistical Analysis 2: Comparison: Placebo vs AMG 301 420 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.79, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = 0.31, 95% CI 2-sided [-2.01 to 2.63]

5. Secondary Outcome: Change From Baseline in Mean Impact on Everyday Activity Domain Scores as Measured by the Migraine Physical Function Impact Diary (MPFID) Over the Last 4 Weeks of the 12-Week Double-Blind Treatment Period
Description: Participants complete the MPFID every day during baseline (Days -28 to Day -1) and the 12-week Double Blind Treatment Period. The MPFID has 2 domains, Impact on Everyday Activities (7 items) and Physical Impairment (5 items), and 1 stand-alone global question that provides an assessment of the overall impact of migraine on participants' everyday activities. The recall period for each item is the past 24 hours.
  The Impact on Everyday Activities Domain Score is reported here. A participant's response to the Impact on Everyday Activities 7 items is measured using a 5-point scale, with difficulty measurements ranging from 1 to 5. The sum was rescaled to a 0 to 100 scale, with 0=no difficulty and 100=unable to do (maximum burden). Negative change from baseline values indicate improvement in migraine impact.
Time Frame: Baseline Day -28 to Day -1; Weeks 9-12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 119 | 93 | 86
units on a scale | -3.42 (0.79) | -4.28 (0.89) | -2.86 (0.92)
Statistical Analysis 1: Comparison: Placebo vs AMG 301 210 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.46, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = -0.86, 95% CI 2-sided [-3.15 to 1.44]
Statistical Analysis 2: Comparison: Placebo vs AMG 301 420 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.64, Mixed Models Analysis — 2-sided significance level of 0.05; difference in least square mean = 0.56, 95% CI 2-sided [-1.77 to 2.89]

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4, where:
  Grade 1 = Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL); Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL; Grade 4 = Life-threatening consequences; urgent intervention indicated Grade 5 = Death related to AE.
Time Frame: Day 1 up to Week 30 (12 weeks of double-blind treatment plus 18 weeks follow-up after last dose of investigational product)
Population: The Safety Analysis Set (SAS) consists of all enrolled participants who received >= 1 dose of investigational product (IP). If a participant received the incorrect dose during the entire double-blind treatment period (DBTP), the participant was analyzed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
Participants
  >= 1 TEAE | 90 | 71 | 65
  Severity grade >= 2 | 41 | 43 | 39
  Severity grade >= 3 | 9 | 5 | 8
  Severity grade >= 4 | 0 | 1 | 0
  Serious TEAE | 3 | 1 | 2
  TEAE leading to discontinuation of IP | 3 | 2 | 5
  Fatal TEAE | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Met Hy's Law Criteria at Baseline and On Study
Description: Hy's law predicts potential for drug-related hepatotoxicity. Hy's Law cases have three components:
  * The drug causes hepatocellular injury, generally defined as an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) by 3-fold or greater above the upper limit of normal (ULN).
  * Among participants showing such aminotransferase elevations, they also have elevation of their serum total bilirubin of greater than 2 times the ULN, without findings of cholestasis (defined as serum alkaline phosphatase activity less than 2 times the upper limit of normal).
  * No other reason can be found to explain the combination of increased aminotransferase and serum total bilirubin, such as viral hepatitis, alcohol abuse, ischemia, preexisting liver disease, or another drug capable of causing the observed injury.
Time Frame: Baseline: Day 1 On study: Weeks 4, 6, 12, 20, 28
Population: Safety analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Baseline | 0 | 0 | 0
  On study: number analyzed (Participants) | 136 | 104 | 100
  On study | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With Aminotransferase Test Abnormalities > 3 Times the Upper Limit of Normal (ULN) at Baseline and On Study
Description: Aminotransferase tests included alanine aminotransferase (ALT) and aspartate aminotransferase (AST). Percentage of participants with results that were greater than 3 * ULN for either test are reported.
Time Frame: Baseline: Day 1 On study: Weeks 4, 6, 12, 20, 28
Population: Safety analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Baseline | 0 | 1.9 | 0
  On study: number analyzed (Participants) | 136 | 104 | 100
  On study | 0.7 | 1.9 | 0

9. Secondary Outcome: Percentage of Participants With Total Bilirubin Test Abnormalities > 2 Times the Upper Limit of Normal (ULN) at Baseline and On Study
Description: Percentage of participants with total bilirubin results that were greater than 2 * ULN are reported.
Time Frame: Baseline: Day 1 On study: Weeks 4, 6, 12, 20, 28
Population: Safety analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Baseline | 0 | 0 | 0
  On study: number analyzed (Participants) | 136 | 104 | 100
  On study | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Systolic Blood Pressure (SBP) in Categories by Visit
Description: Participant was expected to be in a supine position (or the most recumbent position possible) in a rested and calm state for at least 5 minutes before blood pressure assessments were conducted. Blood pressure units are millimeters of mercury (mmHg).
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12,16, 20, 24, 28
Population: Safety analysis population of participants with data at that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Day 1 SBP <90 mmHg: number analyzed (Participants) | 110 | 89 | 81
  Day 1 SBP <90 mmHg | 0.9 | 0.0 | 0.0
  Day 1 SBP > 140 mmHg: number analyzed (Participants) | 110 | 89 | 81
  Day 1 SBP > 140 mmHg | 5.5 | 7.9 | 4.9
  Day 1 SBP > 160 mmHg: number analyzed (Participants) | 110 | 89 | 81
  Day 1 SBP > 160 mmHg | 0.9 | 0.0 | 0.0
  Week 2 SBP < 90 mmHg: number analyzed (Participants) | 134 | 102 | 100
  Week 2 SBP < 90 mmHg | 1.5 | 0.0 | 0.0
  Week 2 SBP > 140 mmHg: number analyzed (Participants) | 134 | 102 | 100
  Week 2 SBP > 140 mmHg | 5.2 | 2.9 | 8.0
  Week 2 SBP > 160 mmHg: number analyzed (Participants) | 134 | 102 | 100
  Week 2 SBP > 160 mmHg | 0.0 | 0.0 | 1.0
  Week 4 SBP < 90 mmHg: number analyzed (Participants) | 135 | 100 | 97
  Week 4 SBP < 90 mmHg | 0.0 | 0.0 | 0.0
  Week 4 SBP > 140 mmHg: number analyzed (Participants) | 135 | 100 | 97
  Week 4 SBP > 140 mmHg | 3.0 | 3.0 | 6.2
  Week 4 SBP > 160 mmHg: number analyzed (Participants) | 135 | 100 | 97
  Week 4 SBP > 160 mmHg | 0.7 | 0.0 | 1.0
  Week 6 SBP < 90 mmHg: number analyzed (Participants) | 131 | 97 | 94
  Week 6 SBP < 90 mmHg | 0.8 | 0.0 | 0.0
  Week 6 SBP > 140 mmHg: number analyzed (Participants) | 131 | 97 | 94
  Week 6 SBP > 140 mmHg | 3.1 | 3.1 | 3.2
  Week 6 SBP > 160 mmHg: number analyzed (Participants) | 131 | 97 | 94
  Week 6 SBP > 160 mmHg | 0.0 | 0.0 | 0.0
  Week 8 SBP < 90 mmHg: number analyzed (Participants) | 130 | 92 | 94
  Week 8 SBP < 90 mmHg | 0.0 | 0.0 | 0.0
  Week 8 SBP > 140 mmHg: number analyzed (Participants) | 130 | 92 | 94
  Week 8 SBP > 140 mmHg | 2.3 | 5.4 | 8.5
  Week 8 SBP > 160 mmHg: number analyzed (Participants) | 130 | 92 | 94
  Week 8 SBP > 160 mmHg | 0.0 | 0.0 | 1.1
  Week 10 SBP < 90 mmHg: number analyzed (Participants) | 122 | 93 | 91
  Week 10 SBP < 90 mmHg | 0.0 | 0.0 | 0.0
  Week 10 SBP > 140 mmHg: number analyzed (Participants) | 122 | 93 | 91
  Week 10 SBP > 140 mmHg | 4.1 | 1.1 | 2.2
  Week 10 SBP > 160 mmHg: number analyzed (Participants) | 122 | 93 | 91
  Week 10 SBP > 160 mmHg | 0.0 | 0.0 | 2.2
  Week 12 SBP < 90 mmHg: number analyzed (Participants) | 125 | 92 | 88
  Week 12 SBP < 90 mmHg | 0.8 | 0.0 | 0.0
  Week 12 SBP > 140 mmHg: number analyzed (Participants) | 125 | 92 | 88
  Week 12 SBP > 140 mmHg | 6.4 | 2.2 | 5.7
  Week 12 SBP > 160 mmHg: number analyzed (Participants) | 125 | 92 | 88
  Week 12 SBP > 160 mmHg | 0.0 | 0.0 | 0.0
  Week 16 SBP < 90 mmHg: number analyzed (Participants) | 113 | 90 | 88
  Week 16 SBP < 90 mmHg | 0.9 | 0.0 | 0.0
  Week 16 SBP > 140 mmHg: number analyzed (Participants) | 113 | 90 | 88
  Week 16 SBP > 140 mmHg | 4.4 | 4.4 | 5.7
  Week 16 SBP > 160 mmHg: number analyzed (Participants) | 113 | 90 | 88
  Week 16 SBP > 160 mmHg | 0.0 | 0.0 | 3.4
  Week 20 SBP < 90 mmHg: number analyzed (Participants) | 113 | 86 | 82
  Week 20 SBP < 90 mmHg | 0.9 | 0.0 | 0.0
  Week 20 SBP > 140 mmHg: number analyzed (Participants) | 113 | 86 | 82
  Week 20 SBP > 140 mmHg | 4.4 | 8.1 | 7.3
  Week 20 SBP > 160 mmHg: number analyzed (Participants) | 113 | 86 | 82
  Week 20 SBP > 160 mmHg | 0.9 | 0.0 | 0.0
  Week 24 SBP < 90 mmHg: number analyzed (Participants) | 106 | 82 | 79
  Week 24 SBP < 90 mmHg | 0.0 | 1.2 | 0.0
  Week 24 SBP > 140 mmHg: number analyzed (Participants) | 106 | 82 | 79
  Week 24 SBP > 140 mmHg | 4.7 | 6.1 | 8.9
  Week 24 SBP > 160 mmHg: number analyzed (Participants) | 106 | 82 | 79
  Week 24 SBP > 160 mmHg | 0.0 | 0.0 | 0.0
  Week 28 SBP < 90 mmHg: number analyzed (Participants) | 108 | 85 | 80
  Week 28 SBP < 90 mmHg | 0.9 | 1.2 | 0.0
  Week 28 SBP > 140 mmHg: number analyzed (Participants) | 108 | 85 | 80
  Week 28 SBP > 140 mmHg | 8.3 | 4.7 | 6.3
  Week 28 SBP > 160 mmHg: number analyzed (Participants) | 108 | 85 | 80
  Week 28 SBP > 160 mmHg | 0.9 | 1.2 | 0.0

11. Secondary Outcome: Percentage of Participants With Diastolic Blood Pressure (DBP) in Categories by Visit
Description: as for outcome 10
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12,16, 20, 24, 28
Population: Safety analysis population of participants with data at that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Day 1 DBP <50 mmHg: number analyzed (Participants) | 110 | 89 | 81
  Day 1 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Day 1 DBP > 90 mmHg: number analyzed (Participants) | 110 | 89 | 81
  Day 1 DBP > 90 mmHg | 4.5 | 6.7 | 7.4
  Day 1 DBP > 100 mmHg: number analyzed (Participants) | 110 | 89 | 81
  Day 1 DBP > 100 mmHg | 0.0 | 1.1 | 0.0
  Week 2 DBP <50 mmHg: number analyzed (Participants) | 134 | 102 | 100
  Week 2 DBP <50 mmHg | 0.7 | 0.0 | 0.0
  Week 2 DBP > 90 mmHg: number analyzed (Participants) | 134 | 102 | 100
  Week 2 DBP > 90 mmHg | 3.7 | 4.9 | 11.0
  Week 2 DBP > 100 mmHg: number analyzed (Participants) | 134 | 102 | 100
  Week 2 DBP > 100 mmHg | 0.7 | 1.0 | 0.0
  Week 4 DBP <50 mmHg: number analyzed (Participants) | 135 | 100 | 97
  Week 4 DBP <50 mmHg | 0.7 | 0.0 | 0.0
  Week 4 DBP > 90 mmHg: number analyzed (Participants) | 135 | 100 | 97
  Week 4 DBP > 90 mmHg | 5.2 | 7.0 | 9.3
  Week 4 DBP > 100 mmHg: number analyzed (Participants) | 135 | 100 | 97
  Week 4 DBP > 100 mmHg | 0.7 | 2.0 | 1.0
  Week 6 DBP <50 mmHg: number analyzed (Participants) | 131 | 97 | 94
  Week 6 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 6 DBP > 90 mmHg: number analyzed (Participants) | 131 | 97 | 94
  Week 6 DBP > 90 mmHg | 9.2 | 3.1 | 7.4
  Week 6 DBP > 100 mmHg: number analyzed (Participants) | 131 | 97 | 94
  Week 6 DBP > 100 mmHg | 0.0 | 0.0 | 1.1
  Week 8 DBP <50 mmHg: number analyzed (Participants) | 130 | 92 | 94
  Week 8 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 8 DBP > 90 mmHg: number analyzed (Participants) | 130 | 92 | 94
  Week 8 DBP > 90 mmHg | 4.6 | 6.5 | 9.6
  Week 8 DBP > 100 mmHg: number analyzed (Participants) | 130 | 92 | 94
  Week 8 DBP > 100 mmHg | 0.0 | 1.1 | 0.0
  Week 10 DBP <50 mmHg: number analyzed (Participants) | 122 | 93 | 91
  Week 10 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 10 DBP > 90 mmHg: number analyzed (Participants) | 122 | 93 | 91
  Week 10 DBP > 90 mmHg | 6.6 | 4.3 | 9.9
  Week 10 DBP > 100 mmHg: number analyzed (Participants) | 122 | 93 | 91
  Week 10 DBP > 100 mmHg | 0.0 | 0.0 | 1.1
  Week 12 DBP <50 mmHg: number analyzed (Participants) | 125 | 92 | 88
  Week 12 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 12 DBP > 90 mmHg: number analyzed (Participants) | 125 | 92 | 88
  Week 12 DBP > 90 mmHg | 7.2 | 3.3 | 8.0
  Week 12 DBP > 100 mmHg: number analyzed (Participants) | 125 | 92 | 88
  Week 12 DBP > 100 mmHg | 0.0 | 0.0 | 1.1
  Week 16 DBP <50 mmHg: number analyzed (Participants) | 113 | 90 | 88
  Week 16 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 16 DBP > 90 mmHg: number analyzed (Participants) | 113 | 90 | 88
  Week 16 DBP > 90 mmHg | 5.3 | 5.6 | 12.5
  Week 16 DBP > 100 mmHg: number analyzed (Participants) | 113 | 90 | 88
  Week 16 DBP > 100 mmHg | 0.0 | 0.0 | 2.3
  Week 20 DBP <50 mmHg: number analyzed (Participants) | 113 | 86 | 82
  Week 20 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 20 DBP > 90 mmHg: number analyzed (Participants) | 113 | 86 | 82
  Week 20 DBP > 90 mmHg | 8.0 | 8.1 | 7.3
  Week 20 DBP > 100 mmHg: number analyzed (Participants) | 113 | 86 | 82
  Week 20 DBP > 100 mmHg | 0.0 | 1.2 | 1.2
  Week 24 DBP <50 mmHg: number analyzed (Participants) | 106 | 82 | 79
  Week 24 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 24 DBP > 90 mmHg: number analyzed (Participants) | 106 | 82 | 79
  Week 24 DBP > 90 mmHg | 4.7 | 7.3 | 11.4
  Week 24 DBP > 100 mmHg: number analyzed (Participants) | 106 | 82 | 79
  Week 24 DBP > 100 mmHg | 0.0 | 2.4 | 1.3
  Week 28 DBP <50 mmHg: number analyzed (Participants) | 108 | 85 | 80
  Week 28 DBP <50 mmHg | 0.0 | 0.0 | 0.0
  Week 28 DBP > 90 mmHg: number analyzed (Participants) | 108 | 85 | 80
  Week 28 DBP > 90 mmHg | 4.6 | 10.6 | 10.0
  Week 28 DBP > 100 mmHg: number analyzed (Participants) | 108 | 85 | 80
  Week 28 DBP > 100 mmHg | 0.0 | 1.2 | 1.3

12. Secondary Outcome: Percentage of Participants With Pulse Rate in Categories by Visit
Description: Participant was expected to be in a supine position (or the most recumbent position possible) in a rested and calm state for at least 5 minutes before pulse assessments were conducted. Pulse rate units are beats per minute (BPM)
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12,16, 20, 24, 28
Population: Safety analysis population of participants with data at that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Day 1 Pulse rate <60 bpm: number analyzed (Participants) | 110 | 89 | 81
  Day 1 Pulse rate <60 bpm | 15.5 | 13.5 | 6.2
  Day 1 Pulse rate >100 bpm: number analyzed (Participants) | 110 | 89 | 81
  Day 1 Pulse rate >100 bpm | 0.0 | 0.0 | 0.0
  Week 2 Pulse rate <60 bpm: number analyzed (Participants) | 134 | 102 | 100
  Week 2 Pulse rate <60 bpm | 11.2 | 4.9 | 6.0
  Week 2 Pulse rate >100 bpm: number analyzed (Participants) | 134 | 102 | 100
  Week 2 Pulse rate >100 bpm | 0.7 | 1.0 | 0.0
  Week 4 Pulse rate <60 bpm: number analyzed (Participants) | 135 | 100 | 97
  Week 4 Pulse rate <60 bpm | 10.4 | 8.0 | 6.2
  Week 4 Pulse rate >100 bpm: number analyzed (Participants) | 135 | 100 | 97
  Week 4 Pulse rate >100 bpm | 0.7 | 0.0 | 0.0
  Week 6 Pulse rate <60 bpm: number analyzed (Participants) | 131 | 97 | 94
  Week 6 Pulse rate <60 bpm | 6.9 | 8.2 | 9.6
  Week 6 Pulse rate >100 bpm: number analyzed (Participants) | 131 | 97 | 94
  Week 6 Pulse rate >100 bpm | 0.8 | 0.0 | 1.1
  Week 8 Pulse rate <60 bpm: number analyzed (Participants) | 130 | 92 | 94
  Week 8 Pulse rate <60 bpm | 9.2 | 7.6 | 12.8
  Week 8 Pulse rate >100 bpm: number analyzed (Participants) | 130 | 92 | 94
  Week 8 Pulse rate >100 bpm | 1.5 | 0.0 | 0.0
  Week 10 Pulse rate <60 bpm: number analyzed (Participants) | 122 | 93 | 91
  Week 10 Pulse rate <60 bpm | 11.5 | 8.6 | 6.6
  Week 10 Pulse rate >100 bpm: number analyzed (Participants) | 122 | 93 | 91
  Week 10 Pulse rate >100 bpm | 0.0 | 0.0 | 0.0
  Week 12 Pulse rate <60 bpm: number analyzed (Participants) | 125 | 92 | 88
  Week 12 Pulse rate <60 bpm | 13.6 | 13.0 | 8.0
  Week 12 Pulse rate >100 bpm: number analyzed (Participants) | 125 | 92 | 88
  Week 12 Pulse rate >100 bpm | 0.0 | 1.1 | 1.1
  Week 16 Pulse rate <60 bpm: number analyzed (Participants) | 113 | 90 | 88
  Week 16 Pulse rate <60 bpm | 10.6 | 8.9 | 8.0
  Week 16 Pulse rate >100 bpm: number analyzed (Participants) | 113 | 90 | 88
  Week 16 Pulse rate >100 bpm | 0.0 | 0.0 | 0.0
  Week 20 Pulse rate <60 bpm: number analyzed (Participants) | 113 | 86 | 82
  Week 20 Pulse rate <60 bpm | 10.6 | 9.3 | 9.8
  Week 20 Pulse rate >100 bpm: number analyzed (Participants) | 113 | 86 | 82
  Week 20 Pulse rate >100 bpm | 0.9 | 1.2 | 1.2
  Week 24 Pulse rate <60 bpm: number analyzed (Participants) | 106 | 82 | 79
  Week 24 Pulse rate <60 bpm | 10.4 | 8.5 | 7.6
  Week 24 Pulse rate >100 bpm: number analyzed (Participants) | 106 | 82 | 79
  Week 24 Pulse rate >100 bpm | 0.0 | 1.2 | 1.3
  Week 28 Pulse rate <60 bpm: number analyzed (Participants) | 108 | 85 | 80
  Week 28 Pulse rate <60 bpm | 8.3 | 11.8 | 10.0
  Week 28 Pulse rate >100 bpm: number analyzed (Participants) | 108 | 85 | 80
  Week 28 Pulse rate >100 bpm | 0.9 | 1.2 | 0.0

13. Secondary Outcome: Percentage of Participants With Temperature in Categories by Visit
Description: Participant was expected to be in a supine position (or the most recumbent position possible) in a rested and calm state for at least 5 minutes before vital sign assessments were conducted. Temperature units are reported in degrees Celsius (C).
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12,16, 20, 24, 28
Population: Safety analysis population of participants with data at that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Day 1 Temperature < 36 C: number analyzed (Participants) | 110 | 89 | 81
  Day 1 Temperature < 36 C | 5.5 | 10.1 | 7.4
  Day 1 Temperature > 38 C: number analyzed (Participants) | 110 | 89 | 81
  Day 1 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 2 Temperature < 36 C: number analyzed (Participants) | 134 | 102 | 100
  Week 2 Temperature < 36 C | 11.2 | 9.8 | 8.0
  Week 2 Temperature > 38 C: number analyzed (Participants) | 134 | 102 | 100
  Week 2 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 4 Temperature < 36 C: number analyzed (Participants) | 135 | 100 | 97
  Week 4 Temperature < 36 C | 8.9 | 12.0 | 10.3
  Week 4 Temperature > 38 C: number analyzed (Participants) | 135 | 100 | 97
  Week 4 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 6 Temperature < 36 C: number analyzed (Participants) | 131 | 97 | 94
  Week 6 Temperature < 36 C | 6.1 | 12.4 | 8.5
  Week 6 Temperature > 38 C: number analyzed (Participants) | 131 | 97 | 94
  Week 6 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 8 Temperature < 36 C: number analyzed (Participants) | 130 | 92 | 94
  Week 8 Temperature < 36 C | 7.7 | 7.6 | 8.5
  Week 8 Temperature > 38 C: number analyzed (Participants) | 130 | 92 | 94
  Week 8 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 10 Temperature < 36 C: number analyzed (Participants) | 122 | 93 | 91
  Week 10 Temperature < 36 C | 9.0 | 14.0 | 7.7
  Week 10 Temperature > 38 C: number analyzed (Participants) | 122 | 93 | 91
  Week 10 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 12 Temperature < 36 C: number analyzed (Participants) | 125 | 92 | 88
  Week 12 Temperature < 36 C | 8.0 | 13.0 | 12.5
  Week 12 Temperature > 38 C: number analyzed (Participants) | 125 | 92 | 88
  Week 12 Temperature > 38 C | 0.8 | 0.0 | 0.0
  Week 16 Temperature < 36 C: number analyzed (Participants) | 113 | 90 | 88
  Week 16 Temperature < 36 C | 6.2 | 7.8 | 13.6
  Week 16 Temperature > 38 C: number analyzed (Participants) | 113 | 90 | 88
  Week 16 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 20 Temperature < 36 C: number analyzed (Participants) | 113 | 86 | 82
  Week 20 Temperature < 36 C | 10.6 | 7.0 | 9.8
  Week 20 Temperature > 38 C: number analyzed (Participants) | 113 | 86 | 82
  Week 20 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 24 Temperature < 36 C: number analyzed (Participants) | 106 | 82 | 79
  Week 24 Temperature < 36 C | 5.7 | 8.5 | 11.4
  Week 24 Temperature > 38 C: number analyzed (Participants) | 106 | 82 | 79
  Week 24 Temperature > 38 C | 0.0 | 0.0 | 0.0
  Week 28 Temperature < 36 C: number analyzed (Participants) | 108 | 85 | 80
  Week 28 Temperature < 36 C | 6.5 | 9.4 | 11.3
  Week 28 Temperature > 38 C: number analyzed (Participants) | 108 | 85 | 80
  Week 28 Temperature > 38 C | 0.0 | 0.0 | 0.0

14. Secondary Outcome: Percentage of Participants With Respiratory Rates in Categories by Visit
Description: Participant was expected to be in a supine position (or the most recumbent position possible) in a rested and calm state for at least 5 minutes before vital sign assessments were conducted. Respiratory rate (RR) is reported in breaths/minute.
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12,16, 20, 24, 28
Population: Safety analysis population of participants with data at that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
Number analyzed (Participants) | 137 | 104 | 102
percentage of participants
  Day 1 RR < 12 breaths/min: number analyzed (Participants) | 108 | 89 | 80
  Day 1 RR < 12 breaths/min | 4.6 | 2.2 | 3.8
  Day 1 RR > 20 breaths/min: number analyzed (Participants) | 108 | 89 | 80
  Day 1 RR > 20 breaths/min | 0.0 | 2.2 | 1.3
  Week 2 RR < 12 breaths/min: number analyzed (Participants) | 134 | 102 | 100
  Week 2 RR < 12 breaths/min | 5.2 | 2.9 | 5.0
  Week 2 RR > 20 breaths/min: number analyzed (Participants) | 134 | 102 | 100
  Week 2 RR > 20 breaths/min | 0.0 | 0.0 | 0.0
  Week 4 RR < 12 breaths/min: number analyzed (Participants) | 135 | 100 | 96
  Week 4 RR < 12 breaths/min | 2.2 | 3.0 | 5.2
  Week 4 RR > 20 breaths/min: number analyzed (Participants) | 135 | 100 | 96
  Week 4 RR > 20 breaths/min | 0.0 | 0.0 | 2.1
  Week 6 RR < 12 breaths/min: number analyzed (Participants) | 131 | 97 | 94
  Week 6 RR < 12 breaths/min | 6.1 | 1.0 | 4.3
  Week 6 RR > 20 breaths/min: number analyzed (Participants) | 131 | 97 | 94
  Week 6 RR > 20 breaths/min | 0.8 | 0.0 | 0.0
  Week 8 RR < 12 breaths/min: number analyzed (Participants) | 130 | 92 | 93
  Week 8 RR < 12 breaths/min | 3.1 | 2.2 | 1.1
  Week 8 RR > 20 breaths/min: number analyzed (Participants) | 130 | 92 | 93
  Week 8 RR > 20 breaths/min | 0.0 | 2.2 | 0.0
  Week 10 RR < 12 breaths/min: number analyzed (Participants) | 122 | 93 | 91
  Week 10 RR < 12 breaths/min | 5.7 | 1.1 | 4.4
  Week 10 RR > 20 breaths/min: number analyzed (Participants) | 122 | 93 | 91
  Week 10 RR > 20 breaths/min | 0.0 | 2.2 | 0.0
  Week 12 RR < 12 breaths/min: number analyzed (Participants) | 125 | 92 | 88
  Week 12 RR < 12 breaths/min | 4.0 | 1.1 | 0.0
  Week 12 RR > 20 breaths/min: number analyzed (Participants) | 125 | 92 | 88
  Week 12 RR > 20 breaths/min | 0.0 | 0.0 | 0.0
  Week 16 RR < 12 breaths/min: number analyzed (Participants) | 113 | 90 | 88
  Week 16 RR < 12 breaths/min | 4.4 | 2.2 | 4.5
  Week 16 RR > 20 breaths/min: number analyzed (Participants) | 113 | 90 | 88
  Week 16 RR > 20 breaths/min | 0.0 | 1.1 | 0.0
  Week 20 RR < 12 breaths/min: number analyzed (Participants) | 113 | 86 | 82
  Week 20 RR < 12 breaths/min | 5.3 | 0.0 | 1.2
  Week 20 RR > 20 breaths/min: number analyzed (Participants) | 113 | 86 | 82
  Week 20 RR > 20 breaths/min | 0.0 | 1.2 | 0.0
  Week 24 RR < 12 breaths/min: number analyzed (Participants) | 106 | 82 | 79
  Week 24 RR < 12 breaths/min | 1.9 | 0.0 | 0.0
  Week 24 RR > 20 breaths/min: number analyzed (Participants) | 106 | 82 | 79
  Week 24 RR > 20 breaths/min | 0.0 | 4.9 | 0.0
  Week 28 RR < 12 breaths/min: number analyzed (Participants) | 108 | 85 | 80
  Week 28 RR < 12 breaths/min | 3.7 | 1.2 | 2.5
  Week 28 RR > 20 breaths/min: number analyzed (Participants) | 108 | 85 | 80
  Week 28 RR > 20 breaths/min | 0.9 | 2.4 | 1.3

ADVERSE EVENTS:
Time Frame: All-cause mortality includes time from enrollment (including the 28 days prior to Day 1), 12-week double-blind treatment and 16-week safety follow-up. Serious adverse events and other adverse events include the 12-week double-blind treatment and 16-week safety follow-up.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Placebo | AMG 301 210 mg Q4W | AMG 301 420 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/104 | 0/102
Serious Adverse Events (participants affected / at risk) | 3/137 | 1/104 | 2/102
Other Adverse Events (participants affected / at risk) | 32/137 | 27/104 | 31/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | AMG 301 210 mg Q4W (N=104) | AMG 301 420 mg Q2W (N=102)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | AMG 301 210 mg Q4W (N=104) | AMG 301 420 mg Q2W (N=102)
Constipation (Gastrointestinal disorders) | 0 | 4 | 6
Fatigue (General disorders) | 8 | 5 | 9
Influenza (Infections and infestations) | 5 | 5 | 6
Nasopharyngitis (Infections and infestations) | 13 | 10 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 1
Migraine (Nervous system disorders) | 3 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03238781/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT03238781/SAP_001.pdf